CLINICAL TRIAL: NCT01663818
Title: Tack Optimized Balloon Angioplasty (TOBA) Study for Femoropopliteal Arteries Using the Tack-IT Endovascular Stapler
Brief Title: Tack Optimized Balloon Angioplasty (TOBA) Study
Acronym: TOBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD 0009
Record Dates: First submitted 2012-08-06; First posted 2012-08-13 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental): Treatment with Tack-IT Endovascular Staple
  Interventions: Device: Tack-It Endovascular Stapler

INTERVENTIONS:
Device: Tack-It Endovascular Stapler

SUMMARY:
A multi-center, post-CE Mark study designed to evaluate the performance of the Intact Vascular Tack-IT Endovascular Stapler™ in subjects with vascular flaps (e.g.; post-angioplasty dissection) resulting from percutaneous transluminal balloon angioplasty (PTA) of superficial femoral or popliteal artery(ies).

DETAILED DESCRIPTION:
Intact Vascular intends to conduct a prospective, single arm, multi-center, post-CE Mark study designed to evaluate the performance of the Intact Vascular Tack-IT Endovascular Stapler™ in subjects with vascular flaps (e.g.; post-angioplasty dissection) resulting from percutaneous transluminal balloon angioplasty (PTA) of superficial femoral or popliteal artery(ies).

ELIGIBILITY:
Inclusion Criteria:

* Rutherford clinical category 2, 3 or 4
* ABI less than or equal to 0.90
* Reference vessel diameter is between 2.5mm and 5.5mm
* Target lesion has stenosis greater than or equal to 70% or is occluded
* Target lesion is less than or equal to 10cm in length

Exclusion Criteria:

* Previously implanted stent in the ipsilateral superficial femoral or popliteal artery
* Target treatment area is severly calcified (e.g. circumferential calcification or calcium plaque visible on plain fluoroscopy that extends far more than 5.0cm continuously)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety | 30 days
  Composite of new-onset major device-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — St. Blasius Hospital; Dierk Scheinert, MD, Principal Investigator — Park Hospital, Leipzig
Locations (1):
- Patrick Peeters, MD, Bonheiden, Belgium